CLINICAL TRIAL: NCT07276347
Title: Comprehensive Assessment of Multiple Products (CAMP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-167
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Hyperopia; Myopia
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (13):
- somofilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: somofilcon A lens
- stenfilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: stenfilcon A lens
- fanfilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: fanfilcon A lens
- comfilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: comfilcon A lens
- verofilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: verofilcon A lens
- serafilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: serafilcon A lens
- lehfilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: lehfilcon A lens
- delefilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: delefilcon A lens
- senofilcon A lens daily disposable (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: senofilcon A daily disposable lens
- senofilcon A lens with blue light technology (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: senofilcon A with blue light technology lens
- senofilcon A lens bi-weekly replacement (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: senofilcon A bi-weekly lens
- samfilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: samfilcon A lens
- kalifilcon A lens (Experimental): Participants will wear thirteen different types of study contact lenses, in a randomized order of testing for the thirteen study contact lens types.
  Interventions: Device: kalilfilcon A lens

INTERVENTIONS:
Device: somofilcon A lens — Participants will be randomized to wear somofilcon A soft contact lens for 10 hours.
  Arms: somofilcon A lens
Device: stenfilcon A lens — Participants will be randomized to wear stenfilcon A soft contact lens for 10 hours.
  Arms: stenfilcon A lens
Device: fanfilcon A lens — Participants will be randomized to wear fanfilcon A soft contact lens for 10 hours.
  Arms: fanfilcon A lens
Device: comfilcon A lens — Participants will be randomized to wear comfilcon A soft contact lens for 10 hours.
  Arms: comfilcon A lens
Device: verofilcon A lens — Participants will be randomized to wear verofilcon A soft contact lens for 10 hours.
  Arms: verofilcon A lens
Device: serafilcon A lens — Participants will be randomized to wear serafilcon A soft contact lens for 10 hours.
  Arms: serafilcon A lens
Device: lehfilcon A lens — Participants will be randomized to wear lehfilcon A soft contact lens for 10 hours.
  Arms: lehfilcon A lens
Device: delefilcon A lens — Participants will be randomized to wear delefilcon A soft contact lens for 10 hours.
  Arms: delefilcon A lens
Device: senofilcon A daily disposable lens — Participants will be randomized to wear senofilcon A soft contact lens for 10 hours.
  Arms: senofilcon A lens daily disposable
Device: senofilcon A with blue light technology lens — Participants will be randomized to wear senofilcon A soft contact lens for 10 hours.
  Arms: senofilcon A lens with blue light technology
Device: senofilcon A bi-weekly lens — Participants will be randomized to wear senofilcon A soft contact lens for 10 hours.
  Arms: senofilcon A lens bi-weekly replacement
Device: samfilcon A lens — Participants will be randomized to wear samfilcon A soft contact lens for 10 hours.
  Arms: samfilcon A lens
Device: kalilfilcon A lens — Participants will be randomized to wear kalifilcon A soft contact lens for 10 hours.
  Arms: kalifilcon A lens

SUMMARY:
The aim of this study is to assess contact lens performance and acceptance.

DETAILED DESCRIPTION:
The objective of this study is to assess the initial performance and acceptance of a range of contact lenses in habitual soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 45 years (inclusive)
2. Habitual soft spherical contact lens wearer (current prescription)
3. Refractive error of -6.00 to -0.50DS or +0.50 to +6.00DS and less than or equal to 0.75DC as vertexed to the corneal plane
4. Anisometropia no greater than 1.50D, based on vertexed manifest refraction spherical equivalent
5. Can achieve visual acuity of at least 20/25 in each eye with spherical equivalent manifest refraction

Exclusion Criteria:

1. Active anterior segment infection, inflammation or abnormality that would contraindicate contact lens wear
2. Use of systemic or ocular medication that would contraindicate contact lens wear
3. Used gas permeable/hard contact lenses (including orthokeratology) in the previous 3 months
4. Participation in a contact lens or lens care product trial in the previous 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
High contrast, high luminance binocular distance visual acuity | At the end of 10 hours of daily wear at dispensing
  High contrast, high luminance binocular distance visual acuity (logMAR) will be measured at 10-hour visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pete Kollbaum, OD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States